CLINICAL TRIAL: NCT06336759
Title: Prospective Clinical Trial Evaluating the Safety and Efficacy of Restylane Lyft and Defyne for Contouring the Jawline
Brief Title: Safety and Efficacy of Fillers for Contouring the Jawline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-10-GAL-JWL
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-03

CONDITIONS: Jawline Contour Deficit
Keywords: Jawline; Injectables; Hyaluronic Acid; Aesthetic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retylane Defyne (Active Comparator): Restylane Defyne is manufactured by Q-Med AB, part of the Galderma Group.
  The product is a sterilized 1ml gel syringe contain 20 mg/mL stabilized HA and 3 mg/mL lidocaine hydrochloride in a physiological buffer (phosphate buffered saline pH 7).
  The participants deemed to have think skin will be treated at the Baseline visit and will be eligible for retreatment 2 weeks later if a touch up is deemed necessary by the Treating Investigator. Volumes used for each subject will be determined by the aesthetic judgement of the Treating Investigator.
  Interventions: Device: Restylane Defyne
- Retylane Lyft (Active Comparator): Restylane Defyne is manufactured by Q-Med AB, part of the Galderma Group.
  The product is a sterilized 1mL gel syringe contain 20 mg/mL stabilized HA and 3 mg/mL lidocaine hydrochloride in a physiological buffer (phosphate buffered saline pH 7).
  The participants deemed to have thick skin will be treated at the Baseline visit and will be eligible for retreatment 2 weeks later if a touch up is deemed necessary by the Treating Investigator. Volumes used for each subject will be determined by the aesthetic judgement of the Treating Investigator.
  Interventions: Device: Restylane Lyft

INTERVENTIONS:
Device: Restylane Defyne — Twenty (20) subjects with thin skin will be recruited and treated with Restylane Defyne.
  Arms: Retylane Defyne
Device: Restylane Lyft — Twenty (20) subjects with thick skin will be recruited and treated with Restylane Lyft.
  Arms: Retylane Lyft

SUMMARY:
The study's goal is to assess the safety and efficacy of two hyaluronic acid products, Restylane Lyft and Defyne, for contouring the jawline and chin, in order to address concerns regarding contour deficiencies among patients seeking aesthetic treatments.

ELIGIBILITY:
Inclusion Criteria:

1. A score > 1 on the Raspaldo Jawline Scale, as assessed by the treating physician at Baseline. A possible secondary deficit of the chin is allowed.
2. Males and females aged > 18 years.
3. Ability to adequately understand the verbal explanations and the written subject information provided in local language and ability and willingness to give consent to participate in the study.
4. Signed and dated informed consent to participate in the study.
5. If female of childbearing potential: a negative urine pregnancy test before all treatments is required.

Exclusion Criteria:

1. Current pregnancy or lactation [sexually active women of childbearing age must agree to use medically acceptable methods of contraception for the duration of this study (e.g., oral contraceptives, condoms, intrauterine device, shot/injection, patch)].
2. Subjects presenting with known allergy to hyaluronic acid fillers or amide local anesthetics.
3. Subjects presenting with porphyria.
4. Subjects with active disease, such as inflammation, infection or tumors, in or near the intended treatment sites.
5. Subjects with history of bleeding disorders or subjects taking thrombolytics or anticoagulants.
6. Subjects taking inhibitors of platelet aggregation (e.g., Aspirin or other non-steroid anti-inflammatory drugs [NSAIDs]), within 2 weeks before treatment.
7. Subjects using immunosuppressants.
8. History of permanent implants in the lower face.
9. History of other treatment/procedure that, in the treating investigator's opinion, would interfere with the study injections and/or study assessments or exposes the subject to undue risk by study participation.
10. Visible markings that in the treating investigator's opinion, may interfere with results or assessments.
11. Inability to comply with follow-up and abstain from other treatments in the region of interest during the study period.
12. Heavy smokers, classified as smoking more than 12 cigarettes per day.
13. History of severe or multiple allergies manifested by anaphylaxis.
14. Previous tissue revitalization therapy in the treatment area within 6 months before treatment with laser or light, mesotherapy, radiofrequency, ultrasound, cryotherapy, chemical peeling, or dermabrasion.
15. Previous treatment with neurotoxins in the area under assessment, within 6 months prior to enrolment.
16. Previous treatment with soft tissue fillers in the area under assessment, within 12 months prior to enrolment.
17. Cancer or precancer in the treatment area (e.g., actinic keratosis).
18. Subjects with a tendency to form hypertrophic scars or any other healing disorders.
19. Subjects with a mean skin thickness in the treatment areas between 1.29mm and 1.49mm (ie, "normal" thickness), as determined by ultrasound at Baseline, to ensure no overlap between the two strata (ie, thin and thick skin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Frequency of subjects having at least "improved" since Baseline, as per the Global Aesthetic Improvement Scale (GAIS) | Baseline to Month 3
  The Global Aesthetic Improvement Scale is a graded Likert scale with assessments ranging form "very much worse" (grade -3) to "very much improved" (grade 3).
Frequency of subjects displaying at least a one grade improvement since Baseline, on the Raspaldo (2008) Jawline Scale | Baseline to Month 3
  The Jawline (Raspaldo 2008) Scale is a 5 point Likert scale ranging from "severe depression or atrophy" (grade 4) to "normal" (grade 1) used by the blinded evaluator to assess the jawline

SECONDARY OUTCOMES:
Frequency of subjects having at least "improved" since Baseline, as per the Global Aesthetic Improvement Scale (GAIS) | Baseline to Month 6
  The Global Aesthetic Improvement Scale is a graded Likert scale with assessments ranging form "very much worse" (grade -3) to "very much improved" (grade 3).
Frequency of subjects displaying at least a one grade improvement since Baseline, on the Raspaldo Jawline Scale | Baseline to Month 6
  The Jawline (Raspaldo 2008) Scale is a 5 point Likert scale ranging from "severe depression or atrophy" (grade 4) to "normal" (grade 1) used by the blinded evaluator to assess the jawline

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nikolis, MD, Principal Investigator — Erevna Innovations Inc.
Locations (1):
- Erevna Innovations Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No